CLINICAL TRIAL: NCT03527589
Title: A Prospective Post Market Study of Patients With Symptomatic Benign Prostatic Hyperplasia Treated by Prostatic Artery Embolization With Embosphere® Microspheres
Brief Title: Embosphere® PROstate Post Market Study
Acronym: PROstate
Status: Completed | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PAE-P4-17-01
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: Prostatic Artery Embolization (PAE); Benign Prostatic Hyperplasia (BPH); Lower Urinary Tract Symptoms (LUTS); Embolization; Embolic; Embosphere Microsphere
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treated with Embosphere Microspheres: Patients with lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH) will be treated with Embosphere Microspheres (size of embolic determined at Investigator discretion).
  Interventions: Device: Prostate artery embolization

INTERVENTIONS:
Device: Prostate artery embolization — Patients with lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH) will be treated with Embosphere Microspheres via prostate artery embolization.

SUMMARY:
Prostatic artery embolization with Embosphere Microspheres is a relatively new procedure. The goal of this post market study is to evaluate long-term safety and effectiveness in a 'real world' setting.

DETAILED DESCRIPTION:
This is a prospective, open label post market study to evaluate the long-term safety and effectiveness of prostatic artery embolization (PAE) using Embosphere Microspheres. Up to 500 patients with lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH) will be enrolled in this single arm post market study. All patients at sites who meet eligibility criteria will be offered participation. Long term effectiveness of PAE on LUTS will be evaluated by International Prostate Symptom Score (IPSS) at baseline, 3 months, 12 months and 24 months. Safety will be assessed by evaluating device or procedure-related adverse events at the same time points, plus at 4 weeks following embolization. Erectile function will be assessed at baseline and 12 months by Sexual Health Inventory for Men (SHIM) score. Additional treatments for refractory or recurrent LUTS due to BPH post prostatic artery embolization will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed informed consent
* Patient age is 18 years or older at time of informed consent
* Patient will undergo prostatic artery embolization with Embosphere Microspheres for the treatment of symptomatic benign prostatic hyperplasia with lower urinary tract symptoms

Exclusion Criteria:

* Patient is unable or unwilling to provide follow-up information
* Patient is undergoing prostatic artery embolization for reasons that do not include symptomatic benign prostatic hyperplasia with lower urinary tract symptoms
* Any other reason the investigator deems cause for exclusion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males can receive prostatic artery embolization
Study Population: Men with lower urinary tract sypmtoms (LUTS) due to benign prostatic hyperplasia (BPH)
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2022-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (8):
  - VA Long Beach Healthcare Systems, Long Beach, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - UC Irvine Health, Orange, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Miami- Miller School of Medicine, Miami, Florida
  - St. Louis University Hospital, St Louis, Missouri
  - Providence Sacred Heart, Spokane, Washington
- Hôspital Européan Georges Pompidou HEGP, Paris, France
- Italy (2):
  - Azienda Ospedaliera S. Croce e Carle Cuneo, Cuneo
  - Ospedale Niguarda Ca' Granda, Milan
- United Kingdom (4):
  - Churchill Hospital, Headington, Oxford
  - Frimley Park Hospital, Camberley, Surrey
  - Royal Bournemouth and Christchurch Hospital, Bournemouth
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sapoval MR, Bhatia S, Dean C, Rampoldi A, Carnevale FC, Bent C, Tapping CR, Bongiovanni S, Taylor J, Brower JS, Rush M, McWilliams JP, Little MW; PROstate Study Investigators. Two-Year Outcomes of Prostatic Artery Embolization for Symptomatic Benign Prostatic Hyperplasia: An International, Multicenter, Prospective Study. Cardiovasc Intervent Radiol. 2024 Nov;47(11):1515-1524. doi: 10.1007/s00270-024-03802-0. Epub 2024 Sep 4. PMID 39230672

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treated With Embosphere Microspheres
Started | 499
Completed | 487
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Treated With Embosphere Microspheres
Number analyzed (Participants) | 487
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 487
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 283
  Unknown or Not Reported | 192
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 332
  More than one race | 0
  Unknown or Not Reported | 147
Region of Enrollment [Number; unit: participants]
  United States | 103
  Italy | 127
  United Kingdom | 122
  France | 135

OUTCOME MEASURES:

1. Primary Outcome: Long-term Effectiveness of Prostatic Artery Embolization (PAE) With Embosphere Microspheres as Assessed by the International Prostate Symptom Score (IPSS).
Description: The two time points used in the calculation were baseline and 12 months. The calculation was done using the 12 months mean International Prostate Symptom Score (IPSS) minus the baseline mean IPSS for paired data (e.g., available data on both baseline and 12 month timepoints). From the IPSS questionnaire, the total score was used and range from 0 to 35 with lower scores representing better outcomes and higher scores representing worse outcomes. There are a total of 7 questions on the scale and the scores from each question are summed to get a total score. A negative change score means improvement of outcomes. 'Scores on a scale' is the unite of measure
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Treated With Embosphere Microspheres
Number analyzed (Participants) | 487
scores on scale | -11.1 [-11.9 to -10.2]

2. Secondary Outcome: International Prostate Symptom Score (IPSS) After Discontinuation of Indwelling Bladder Catheter (IBC) Post PAE.
Description: The time points used in the calculation were baseline, 3 months and 24 months. The calculation was done using the 3 months mean International Prostate Symptom Score (IPSS) minus the baseline mean IPSS for paired data (e.g., available data on both baseline and 3 month timepoints). The same calculation was also done at 24 months. From the IPSS questionnaire, the total score was used and range from 0 to 35 with lower scores representing better outcomes and higher scores representing worse outcomes. There are a total of 7 questions on the scale and the scores from each question are summed to get a total score. A negative change score means improvement of outcomes. 'Scores' on a scale is the unite of measure.
Time Frame: 3, 24 Months
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Treated With Embosphere Microspheres
Number analyzed (Participants) | 487
scores on scale
  3 Months | -12.4 [-13.2 to -11.6]
  24 Months | -10.1 [-11.1 to -9.1]

3. Secondary Outcome: Quality of Life Due to Urinary Symptoms After Discontinuation of Indwelling Bladder Catheter (IBC) Post Prostate Artery Embolization (PAE) Using the International Prostate Symptom Score (IPSS) Quality of Life Assessment Index.
Description: as for outcome 2
Time Frame: 3, 24 Months
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Treated With Embosphere Microspheres
Number analyzed (Participants) | 487
scores on scale
  3 Months | -2.7 [-2.9 to -2.5]
  24 Months | -2.4 [-2.6 to -2.2]

4. Secondary Outcome: Device or Procedure Related Adverse Events Post Procedure.
Description: The measure used to assess "device or procedure related adverse events post procedure" at three different time points (3, 12, 24 months) are frequencies and percentages. For each visit (or reporting time point), the event rate will be calculated as the number of subjects with certain event terms over the number of evaluable subjects. The evaluable subjects at each reporting time point include all subjects who are enrolled and
  1. had an event within (on or before) the reporting cutoff days, or
  2. had a follow-up at or after the lower limit of the reporting window, or
  3. the withdrawal consent date/recorded lost-to-follow-up date at or after the lower limit of the reporting window.
Time Frame: 3, 12, 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Embosphere Microspheres
Number analyzed (Participants) | 487
Participants
  3 Months | 0
  12 Months | 0
  24 Months | 0

5. Secondary Outcome: Frequency of Indwelling Bladder Catheter (IBC) Removal Post PAE.
Time Frame: 3, 12, 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Embosphere Microspheres
Number analyzed (Participants) | 487
Participants
  3 Months | 55
  12 Months | 0
  24 Months | 0

6. Secondary Outcome: Technical Success Defined as Successful Embolization of the Treated Prostate Gland.
Time Frame: Day of PAE Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Embosphere Microspheres
Number analyzed (Participants) | 487
Participants | 432

7. Secondary Outcome: Additional Treatments for Refractory or Recurrent Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH) Post Prostatic Artery Embolization (PAE).
Time Frame: 3, 12, 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Treated With Embosphere Microspheres
Number analyzed (Participants) | 487
Participants
  3 Months | 20
  12 Months | 22
  24 Months | 10

8. Secondary Outcome: Change From Baseline in Erectile Function Post Prostatic Artery Embolization (PAE) Using the Sexual Health Inventory for Men (SHIM).
Description: The calculation was done using the 12 months mean Sexual Health Inventory for Men (SHIM) score minus the baseline mean SHIM score for paired data (e.g., available data on both baseline and 12 month timepoints). From the SHIM questionnaire, the total scores was used and range from 1 to 25 with higher scores representing better outcomes (no signs of erectile dysfunction) and lower scores representing worse outcomes (severe erectile dysfunction). There are a total of 5 questions on the scale and the scores from each question are summed to get a total score. A positive change score means improvement of outcomes. 'Scores' on a scale is the unite of measure.
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Treated With Embosphere Microspheres
Number analyzed (Participants) | 487
scores on scale | -0.1 [-0.8 to 0.6]

ADVERSE EVENTS:
Time Frame: 24 Months
Description: Results in death Is life-threatening Requires in-patient hospitalization or prolongation of existing hospitalization Results in persistent or significant disability/incapacity Is a congenital anomaly/birth defect Is an important medical event
Arm/Group | Treated With Embosphere Microspheres
All-Cause Mortality (participants affected / at risk) | 0/487
Serious Adverse Events (participants affected / at risk) | 10/487
Other Adverse Events (participants affected / at risk) | 57/487
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated With Embosphere Microspheres (N=487)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Blood in urine (Renal and urinary disorders) | 1 (1)
Dizziness upon walking (General disorders) | 1 (1)
Dyspnea and congestive heart failure (Cardiac disorders) | 1 (1)
Emergency admission with abdominal pain and vomiting (General disorders) | 1 (1)
False aneurysm at point of puncture (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Prostatitis (Infections and infestations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection and hypotension (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated With Embosphere Microspheres (N=487)
Abdominal spasm (Gastrointestinal disorders) | 5 (6)
Acute retention of urine (Gastrointestinal disorders) | 2 (2)
Blood in stool (Gastrointestinal disorders) | 3 (3)
Bowel incontinence (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 20 (20)
Fever (General disorders) | 1 (1)
Low Grade Fever (Gastrointestinal disorders) | 1 (1)
Pain (Gastrointestinal disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Post procedural pain (Injury, poisoning and procedural complications) | 4 (4)
Burning sensation (Nervous system disorders) | 2 (2)
Bladder inability to empty (Renal and urinary disorders) | 4 (4)
Bladder spasm (Renal and urinary disorders) | 6 (7)
Burning micturition (Renal and urinary disorders) | 29 (30)
Contracted bladder (Renal and urinary disorders) | 1 (1)
Frequency urinary (Renal and urinary disorders) | 12 (13)
Hematuria (Renal and urinary disorders) | 14 (14)
Incontinence urinary (Renal and urinary disorders) | 9 (10)
Painful urination (Renal and urinary disorders) | 31 (32)
Unable to urinate (Renal and urinary disorders) | 2 (2)
Urgency urination (Renal and urinary disorders) | 10 (11)
Urinary catheterization (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 2 (2)
Bloody semen (Reproductive system and breast disorders) | 11 (11)
Pelvic pain (Reproductive system and breast disorders) | 13 (13)
Penile pain (Reproductive system and breast disorders) | 1 (2)
Rectoprostatic fistula (Reproductive system and breast disorders) | 1 (1)
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03527589/Prot_SAP_000.pdf